CLINICAL TRIAL: NCT04894864
Title: Effect of a Perioperative Opioid Free Anesthesia-Analgesia (OFA-A) Strategy on Surgical Stress Response in Elective Open Abdominal Aortic Aneurysm Repair: A Prospective Randomized Study
Brief Title: Opioid Free Anesthesia-Analgesia Strategy and Surgical Stress in Elective Open Abdominal Aortic Aneurysm Repair
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Crete (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, George Papastratigakis, MD, Principal Investigator, University of Crete
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OFA-aneurysm
Record Dates: First submitted 2021-04-19; First posted 2021-05-20 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Elective Surgical Procedures; Postoperative Pain; Anesthesia; Opioid Use; Abdominal Aortic Aneurysm Without Rupture; Vascular Surgical Procedure; Interleukin 6; Immunomodulators
Keywords: Opioid-free Anesthesia-Analgesia; Cytokines; Opioid-based Anesthesia-Analgesia; Haemodynamic Stability; Open Abdominal Aortic Aneurysm Repair; Immunomodulation; Inflammatory Markers
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Implementation of a multimodal anesthetic opioid-free strategy, that includes the administration of pregabalin, ketamine, dexmedetomidine, lidocaine, dexamethasone, magnesium sulphate, paracetamol and dexketoprofen is anticipated to modulate the inflammatory and stress response, as measured by levels of inflammatory markers and haemodynamic stability, compared to conventional anesthetic opioid-based techniques. Furthermore, a decreased inflammatory and stress response, as expressed by reduced levels of inflammatory biomarkers and hemodynamic stability, is expected to decrease peripheral and central sensitization, contributing to better postoperative analgesia.
Who Masked: Participant, Investigator
Masking Description: Laboratory data analysis collaborators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid-Based Anesthesia Analgesia (Active Comparator): Premedication: IM Midazolam 0.05-0.07mg/kg. Anesthesia induction: Midazolam 0.03mg/kg, Propofol 2-3mg/kg, Fentanyl 1-2mcg/kg and Cisatracurium 0.2mg/kg or alternatively Rocuronium 0.6-1.2mg/kg. Anesthesia maintenance: Desflurane set at approximately 1 MAC, Morphine 0.1-0.12mg/kg, Fentanyl 1-2mcg/kg during induction and 50-100mcg prn, Paracetamol 1g +/- Dexketoprofen trometamol 50mg, along with Ondansetron 4mg or Droperidol 0.625mg. Wound infiltration: Ropivacaine 75-150mg. ICU stay sedation: Remifentanil infusion, until removal of the endotracheal tube. Surgical ward: PCA pump with Morphine for the first 3 postoperative days. Additional postoperative analgesia: Paracetamol 1g x3 +/- Dexketoprofen trometamol 50mg x2. Rescue therapy only: Tramadol 50-100mg.
  Interventions: Drug: Opioid-Based Anesthesia-Analgesia Strategy
- Opioid-Free Anesthesia Analgesia (Active Comparator): Premedication: Pregabalin 50-150mg x2, IM Midazolam 0.05-0.07mg/kg. Anesthesia induction: Midazolam 0.03mg/kg, Dexdmedetomidine 0.5-1mcg/kg, Lidocaine 1mg/kg, Propofol 2-3mg/kg, Ketamine 1-1.5mg/kg, Hyoscine 10mg, Cisatracurium 0.2mg/kg or alternatively Rocuronium 0.6-1.2mg/kg, Magnesium sulphate 2.5-5g and Dexamethasone 8-16mg. Anesthesia maintenance: Desflurane set at ~1 MAC, Dexmedetomidine 0.2-1.2mcg/kg/h, Lidocaine 0.5-1mg/kg/h, Ketamine 0.3-0.5mg/kg prn, Paracetamol 1g +/- Dexketoprofen trometamol 50mg, and Ondansetron 4mg or Droperidol 0.625mg. Wound infiltration: Ropivacaine 75-150mg. ICU sedation: Dexmedetomidine + Lidocaine infusions, until removal of the ETT. Surgical ward: PCA pump with Ketamine, Lidocaine, Clonidine and Midazolam for the first 3 postoperative days. Additionally, Pregabalin 50mg per os x1 and 25mg x1, up to x2, Paracetamol 1g x3 +/- Dexketoprofen trometamol 50mg x2. Rescue therapy only: Tramadol 50-100mg.
  Interventions: Drug: Opioid-free Anesthesia-Analgesia Strategy

INTERVENTIONS:
Drug: Opioid-Based Anesthesia-Analgesia Strategy — A perioperative Opioid-Based multimodal Anesthesia-Analgesia strategy will be implemented as described in the Opioid-Based arm of the study.
  Other Names: Opioid-Based Anesthesia; OBA-A
  Arms: Opioid-Based Anesthesia Analgesia
Drug: Opioid-free Anesthesia-Analgesia Strategy — A perioperative Opioid-Free multimodal Anesthesia-Analgesia strategy will be implemented as described in the Opioid-Free arm of the study.
  Other Names: Opioid-Free Anesthesia; OFA-A
  Arms: Opioid-Free Anesthesia Analgesia

SUMMARY:
Open Abdominal Aortic Aneurysm (AAA) repair is a high-risk surgical procedure accompanied by intense endocrine and metabolic responses to surgical stress, with subsequent activation of the inflammatory cascade, cytokine and acute-phase protein release, and bone marrow activation. There is a proven correlation of surgical stress, which patients undergoing open AAA repair are subjected to, with patient outcome, morbidity/mortality, intensive care unit stay and overall length of stay. Modern general anesthetic techniques have been revised and rely on perioperative multimodal anesthetic and analgesic strategies for improved overall patient outcome. Based on this context of a multimodal anesthetic technique and having taken into consideration the international "opioid-crisis" epidemic, an Opioid Free Anesthesia-Analgesia (OFA-A) strategy started to emerge. It is based on the administration of a variety of anesthetic/analgesic agents with different mechanisms of action, including immunomodulating and anti-inflammatory effects.

Our basic hypothesis is that the implementation of a perioperative multimodal OFA-A strategy, involving the administration of pregabalin, ketamine, dexmedetomidine, lidocaine, dexamethasone, dexketoprofen, paracetamol and magnesium sulphate, will lead to attenuation of surgical stress response compared to a conventional Opioid-Based Anesthesia-Analgesia (OBA-A) strategy. Furthermore, the anticipated attenuation of the inflammatory response, is pressumed to be associated with equal or improved analgesia, compared to a perioperative OBA-A technique.

DETAILED DESCRIPTION:
Open abdominal aortic aneurysm (AAA) repair surgery is a high-risk operation, often performed on high-risk patients. Despite advancements made in diagnosis, management, surgical techniques and treatment of these patients, morbidity and mortality remain high. Mortality after open AAA repair remains higher than the average mortality of the matched population for age and sex. Debate is ongoing as to whether open AAA repair or endovascular aneurysm repair (EVAR) is better in terms of overall long-term survival rate.

Regarding open AAA repair, the very nature of the surgery itself, with surgical trauma, aortic cross clamping and its resulting ischemia-reperfusion injury, and cellular interactions of blood with the biomaterial surface of the graft, causes intense and varied metabolic, endocrine and immunological responses. These surgical stress-related responses are evident as marked increases in inflammatory cytokines such as TNF-a, IL-1a, IL-6, IL-8, IL-10, stimulation of the sympathetic system, and stimulation of the hypothalamic-pituitary-adrenal axis, caused by release of CRH and AVP. High levels of IL-6, peaking at 4-48h after clamp removal, have been associated with serious postoperative complications and its levels reflect the intensity of surgical trauma following AAA repair. Other inflammation markers such as CRP and leukocytes have also been shown to increase postoperatively.

While the surgical technique has been extensively studied as to the role it plays on the control of the surgical stress response, patient outcome, morbidity and overall mortality, fewer studies have been conducted to study the effect of the anesthetic management on these factors. While most of them have been focusing on the comparison of general anesthetic vs regional techniques, only few compare different general anesthetic techniques on patient outcome.

Modern general anesthetic techniques have been revised and rely on a multimodal anesthetic and analgesic perioperative regimen for improved patient outcome. A multimodal regimen requires the administration of at least 2 factors with different mechanisms of action. At least one factor causes inhibition of central sensitization and at least another one inhibits the peripheral sensitization of the nervous system, as a response to painful surgical stimuli, mitigating adverse neuroplasticity. One such example, is an Opioid-Free Anesthetic-Analgesic (OFA-A) strategy, which implements a variety of pharmacological agents, including some with demonstrated immunomodulating and anti-inflammatory effects. Apart from sparing any opioid-related adverse effects, an OFA-A multimodal strategy targets optimal analgesia with a multitude of factors in the lowest possible dose, aiming for additive or synergistic effects. An additional advantage of using an OFA-A technique is the prevention of opioid-induced hyperalgesia.

Our hypothesis is that implementation of a multimodal OFA-A strategy, leads to a decreased sympathetic and inflammatory response, compared to conventional opioid-based anesthetic techniques. A decreased inflammatory and stress response as expressed by reduced levels of IL-6, IL-8, IL-10, TNF-a, CRP, cortisol, arginine vasopressin (AVP), white blood cells count and hemodynamic stability is expected to decrease peripheral and central sensitization, contributing to better postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Consent
2. Age between 40 and 85 years old
3. Patients undergoing Elective Open Abdominal Aortic Infrarenal Aneurysm Repair

Exclusion Criteria:

1. Immunocompromised patients
2. Patients with active infection
3. Reoperation on the aorta
4. Inflammatory bowel Disease
5. Malignancy
6. Chronic Inflammatory conditions (e.g. Rheymatoid arthritis, Psoriatic arthritis)
7. Chronic corticosteroid or immunosuppressive drug use
8. Intraoperative transfusion with >2 units of packed Red Blood Cells

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
Surgical Stress Response - IL-6 - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by IL-6 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-6 - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by IL-6 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-6 - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by IL-6 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-6 - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by IL-6 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-8 - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by IL-8 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-8 - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by IL-8 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-8 - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by IL-8 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-8 - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by IL-8 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-10 - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by IL-10 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-10 - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by IL-10 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-10 - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by IL-10 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - IL-10 - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by IL-10 serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - AVP - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by AVP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - AVP - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by AVP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - AVP - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by AVP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - AVP - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by AVP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - TNF-a - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by TNF-a serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - TNF-a - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by TNF-a serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - TNF-a - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by TNF-a serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - TNF-a - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by TNF-a serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - Cortisol - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by cortisol serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - Cortisol - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by cortisol serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - Cortisol - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by cortisol serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - Cortisol - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by cortisol serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - CRP - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by CRP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - CRP - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by CRP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - CRP - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by CRP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - CRP - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by CRP serum levels. Blood sample collection will take place in both study groups.
Surgical Stress Response - WBC - Preoperatively | 1) Preoperatively (as a baseline)
  Inflammatory response and stress response as quantified by WBC count. Blood sample collection will take place in both study groups.
Surgical Stress Response - WBC - 15 minutes after aortic cross-clamp | 2) 15 minutes after aortic cross-clamping
  Inflammatory response and stress response as quantified by WBC count. Blood sample collection will take place in both study groups.
Surgical Stress Response - WBC - 60 minutes after aortic cross-clamp | 3) 60 minutes after aortic cross-clamp release
  Inflammatory response and stress response as quantified by WBC count. Blood sample collection will take place in both study groups.
Surgical Stress Response - WBC - 24 hours after aortic cross-clamp release | 4) 24 hours after aortic cross-clamp release
  Inflammatory response and stress response as quantified by WBC count. Blood sample collection will take place in both study groups.
Haemodynamic Stability - Coefficient of Variation PR | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Rate - PR. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. The Coefficient of variation of the PR values will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Average Real Variability PR | Every minute from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Average Real Variability of the PR. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Values will be averaged every minute and the Average Real Variability will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Coefficient of Variation SBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Systolic Blood Pressure - SBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. The Coefficient of variation of SBP values will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Average Real Variability SBP | Every minute from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Average Real Variability of the SBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Values will be averaged every minute and the Average Real Variability will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Coefficient of Variation DBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Diastolic Blood Pressure - DBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. The Coefficient of variation of DBP values will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Average Real Variability DBP | Every minute from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Average Real Variability of the DBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Values will be averaged every minute and the Average Real Variability will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Coefficient of Variation MBP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Mean Blood Pressure - MBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. The Coefficient of variation of MBP values will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Average Real Variability MBP | Every minute from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Average Real Variability of the MBP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Values will be averaged every minute and the Average Real Variability will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Coefficient of Variation PP | Every 20 seconds from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Pulse Pressure. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. The Coefficient of variation of PP values will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Average Real Variability PP | Every minute from anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours.
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Average Real Variability of the PP. Data will be collected from a pulse contour analysis monitor, and values will be collected every 20 seconds. Values will be averaged every minute and the Average Real Variability will be reported for each patient, extracted from the collected data.
Haemodynamic Stability - Tachycardia | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Intraoperative Tachycardia (defined as PR≥ 100 bpm), with episodes lasting ≥1 minute. Data will be reported in as a percentage of the total surgical time in which the participant exhibited tachycardia.
Haemodynamic Stability - Bradycardia | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Intraoperative Bradycardia (defined as PR≤ 40 bpm), with episodes lasting ≥1 minute. Data will be reported in as a percentage of the total surgical time in which the participant exhibited bradycardia.
Haemodynamic Stability - Hypotension SBP | Baseline: 5 minutes prior to anaesthesia induction. Intraoperative Hypotension: From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Intraoperative Hypotension (defined as SBP≤90mmHg or ≤80% of preoperative Baseline), with episodes lasting ≥1 minute. All patients will have a 5 minute preoperative SBP baseline, with measurements every 20 seconds. Intraoperative data will be compared to the mean preoperative 5 minute SPB baseline. Data will be reported in as a percentage of the total surgical time in which the participant exhibited hypotension, based on the SBP values.
Haemodynamic Stability - Hypotension MBP | Baseline: 5 minutes prior to anaesthesia induction. Intraoperative Hypotension: From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Intraoperative Hypotension (defined as MBP≤65mmHg or ≤80% of preoperative Baseline), with episodes lasting ≥1 minute. All patients will have a 5 minute preoperative MBP baseline, with measurements every 20 seconds. Intraoperative data will be compared to the mean preoperative 5 minute MPB baseline. Data will be reported in as a percentage of the total surgical time in which the participant exhibited hypotension, based on the MBP values.
Haemodynamic Stability - Hypertension | Baseline: 5 minutes prior to anaesthesia induction. Intraoperative Hypotension: From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Intraoperative Hypertension (defined as SBP ≥120% of preoperative Baseline), with episodes lasting ≥1 minute. All patients will have a 5 minute preoperative SBP baseline, with measurements every 20 seconds. Intraoperative data will be compared to the mean preoperative 5 minute SPB baseline. Data will be reported in as a percentage of the total surgical time in which the participant exhibited hypertension, based on the SBP values.
Haemodynamic Stability - Fluid requirements - Crystalloids - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Crystaloid Fluid Requirements averaged over the total surgical time. Data will be reported in ml/kg*h.
Haemodynamic Stability - Fluid requirements - Crystalloids - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Crystaloid Fluid Requirements. Data will be reported in ml/kg*h.
Haemodynamic Stability - Fluid requirements - Colloids - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Colloid Fluid Requirements averaged over the total surgical time. Data will be reported in ml/kg*h.
Haemodynamic Stability - Fluid requirements - Colloids - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Colloid Fluid Requirements. Data will be reported in ml/kg*h.
Haemodynamic Stability - Fluid requirements - Concentrated RBCs - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Concentrated RBC unit Requirements. Data will be reported in ml.
Haemodynamic Stability - Fluid requirements - Concentrated RBCs - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Concentrated RBC unit Requirements. Data will be reported in ml.
Haemodynamic Stability - Fluid requirements - Plasma - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Plasma unit Requirements. Data will be reported in ml.
Haemodynamic Stability - Fluid requirements - Plasma - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Plasma unit Requirements. Data will be reported in ml.
Haemodynamic Stability - Fluid requirements - Platelets - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Platelet unit Requirements. Data will be reported in ml.
Haemodynamic Stability - Fluid requirements - Platelets - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Platelet unit Requirements. Data will be reported in ml.
Haemodynamic Stability - Blood Loss - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Blood Loss. Data will be reported in ml.
Haemodynamic Stability - Blood Loss - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Blood Loss. Data will be reported in ml.
Haemodynamic Stability - Fluid Balance - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Fluid Balance averaged over the total surgical time. Data will be reported in ml/kg/h
Haemodynamic Stability - Fluid Balance - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Fluid Balance. Data will be reported in ml.
Haemodynamic Stability - Vasoactive Requirements - Adrenaline - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Adrenaline requirements. Data will be reported in mg.
Haemodynamic Stability - Vasoactive Requirements - Adrenaline - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Adrenaline requirements. Data will be reported in mg.
Haemodynamic Stability - Vasoactive Requirements - Noradrenaline - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Noradrenaline requirements. Data will be reported as an averaged intraoperative rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Noradrenaline - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Noradrenaline requirements. Data will be reported as an averaged rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Ephedrine - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Ephedrine requirements. Data will be reported in mg.
Haemodynamic Stability - Vasoactive Requirements - Ephedrine - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Ephedrine requirements. Data will be reported in mg.
Haemodynamic Stability - Vasoactive Requirements - Phenylephrine - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Phenylephrine requirements. Data will be reported as an averaged intraoperative rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Phenylephrine - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Phenylephrine requirements.Data will be reported as an averaged rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Dobutamine - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Dobutamine requirements. Data will be reported as an averaged intraoperative rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Dobutamine - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Dobutamine requirements. Data will be reported as an averaged rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Dopamine - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Dopamine requirements. Data will be reported as an averaged intraoperative rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Dopamine - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Dopamine requirements. Data will be reported as an averaged rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Nitroglycerine - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Nitroglycerine requirements. Data will be reported as an averaged intraoperative rate in mcg/kg*min.
Haemodynamic Stability - Vasoactive Requirements - Nitroglycerine - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Haemodynamic Stability as quantified by hemodynamic markers, specifically Nitroglycerine requirements. Data will be reported as an averaged rate in mcg/kg*min.

SECONDARY OUTCOMES:
Postoperative pain - Numerical Rating Scale (NRS) - Immediately Postoperatively | 1) Immediately postoperatively (if awakened prior to ICU admission)
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Postoperative pain - Numerical Rating Scale (NRS) - First postoperative day | 2) First postoperative day
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Postoperative pain - Numerical Rating Scale (NRS) - Second postoperative day | 3) Second postoperative day
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Postoperative pain - Numerical Rating Scale (NRS) - Third postoperative day | 4) Third postoperative day
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Postoperative pain - Critical Care Pain Observation Tool (CPOT) - Immediately Postoperatively | 1) Immediately postoperatively (if awakened prior to ICU admission)
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Postoperative pain - Critical Care Pain Observation Tool (CPOT) - First postoperative day | 2) First postoperative day
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Postoperative pain - Critical Care Pain Observation Tool (CPOT) - Second postoperative day | 3) Second postoperative day
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Postoperative pain - Critical Care Pain Observation Tool (CPOT) - Third postoperative day | 4) Third postoperative day
  Evaluation of patients' pain using scales: Critical Care Pain Observation Tool (CPOT). The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients or vocalization for extubated patients. Patient's behavior in each domain is scored between 0 and 2. The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Intolerable - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Intolerable" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Intolerable - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Intolerable" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Intolerable - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Intolerable" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Tolerable with discomfort - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Tolerable with discomfort" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Tolerable with discomfort - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Tolerable with discomfort" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Tolerable with discomfort - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Tolerable with discomfort" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Comfortably manageable - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Comfortably manageable" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Comfortably manageable - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Comfortably manageable" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Comfortably manageable - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Comfortably manageable" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Negligible Pain - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Negligible Pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Negligible Pain - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Negligible Pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Comfort - Negligible Pain - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to how comfortable patients feel with their pain, available answers will be:
  1. Intolerable
  2. Tolerable with discomfort
  3. Comfortably manageable
  4. Negligible Pain
  The percentage of patients that report pain that is "Negligible Pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting Worse - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting worse" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting Worse - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting worse" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting Worse - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting worse" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - About the same - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "About the same" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - About the same - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "About the same" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - About the same - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "About the same" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting better | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting better" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting better - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting better" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Change in Pain - Getting better - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to changes in pain perception by patients, available answers will be:
  1. Getting worse
  2. About the same
  3. Getting better
  The percentage of patients that report pain that is "Getting better" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Inadequate pain control - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Inadequate pain control" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Inadequate pain control - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Inadequate pain control" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Inadequate pain control - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report "Inadequate pain control" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Effective, just about right - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report pain control that is "Effective, just about right" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Effective, just about right - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report pain control that is "Effective, just about right" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Effective, just about right - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients that report pain control that is "Effective, just about right" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Would like to reduce medication - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients whose pain control is reported as "Would like to reduce medication" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Would like to reduce medication - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients whose pain control is reported as "Would like to reduce medication" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Pain control - Would like to reduce medication - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to pain control reported by patients, available answers will be:
  1. Inadequate pain control
  2. Effective, just about right
  3. Would like to reduce medication
  The percentage of patients whose pain control is reported as "Would like to reduce medication" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can't do anything because of pain - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can't do anything because of pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can't do anything because of pain - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can't do anything because of pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can't do anything because of pain - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can't do anything because of pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Pain keeps me from doing most of what I need to do - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Pain keeps me from doing most of what I need to do" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Pain keeps me from doing most of what I need to do - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Pain keeps me from doing most of what I need to do" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Pain keeps me from doing most of what I need to do - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Pain keeps me from doing most of what I need to do" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do most things, but pain gets in the way of some - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do most things, but pain gets in the way of some" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do most things, but pain gets in the way of some - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do most things, but pain gets in the way of some" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do most things, but pain gets in the way of some - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do most things, but pain gets in the way of some" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do everything I need to do - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do everything I need to do" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do everything I need to do - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do everything I need to do" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Functioning - Can do everything I need to do - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to functioning - for the usual things patients need to do, available answers will be:
  1. Can't do anything because of pain
  2. Pain keeps me from doing most of what I need to do
  3. Can do most things, but pain gets in the way of some
  4. Can do everything I need to do
  The percentage of patients whose functioning is reported as "Can do everything I need to do" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with pain most of the night - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with pain most of the night" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with pain most of the night - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with pain most of the night" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with pain most of the night - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with pain most of the night" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with occasional pain - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with occasional pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with occasional pain - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with occasional pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Awake with occasional pain - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Awake with occasional pain" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Normal sleep - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Normal sleep" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Normal sleep - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Normal sleep" will be reported
Postoperative pain - Clinically Aligned Pain Assessment Tool (CAPA) - Sleep - Normal sleep - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain using scales: Clinically Aligned Pain Assessment Tool (CAPA). Patients will be given a standardized CAPA questionaire that has pre-determined answers that patients will be able to choose from, to best describe their pain. In regards to sleep, if the pain is waking patients up, available answers will be:
  1. Awake with pain most of the night
  2. Awake with occasional pain
  3. Normal sleep
  The percentage of patients whose sleep is reported as "Normal sleep" will be reported
Analgesic Requirements - First postoperative day | 1) First postoperative day
  Evaluation of patients' pain by recording the number of times that rescue analgesia (tramadol) was required.
Analgesic Requirements - Second postoperative day | 2) Second postoperative day
  Evaluation of patients' pain by recording the number of times that rescue analgesia (tramadol) was required.
Analgesic Requirements - Third postoperative day | 3) Third postoperative day
  Evaluation of patients' pain by recording the number of times that rescue analgesia (tramadol) was required.
Kidney function - Furosemide requirement - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Kidney function as quantified by furosemide requirement to maintain urine output. Data will be reported in mg.
Kidney function - Furosemide requirement - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Kidney function as quantified by furosemide requirement to maintain urine output. Data will be reported in mg.
Kidney function - MDRD GFR - Preoperatively | 1) Preoperatively (as a baseline)
  Kidney function as assessed by preoperative GFR calculated by the MDRD GFR equation.
Kidney function - MDRD GFR - Immediately postoperatively | 2) At the end of surgery 1h after the end of placement of last suture/surgical clip on patient, upon ICU admission.
  Kidney function as assessed by postoperative GFR calculated by the MDRD GFR equation.
Kidney function - MDRD GFR - 24h Postoperatively | 3) 24h postoperatively
  Kidney function as assessed by postoperative GFR calculated by the MDRD GFR equation.
Kidney function - Urine Output - Intraoperatively | From anesthesia induction, until the end of surgery (end of placement of last suture/surgical clip on patient), assessed up to 8 hours
  Kidney function as quantified by urine output. Data will be reported as an averaged intraoperative rate in ml/kg*h.
Kidney function - Urine Output - 24 hours postoperatively | From the end of surgery (end of placement of last suture/surgical clip on patient) until 24 hours postoperatively
  Kidney function as quantified by urine output. Data will be reported as an averaged rate in ml/kg*h.
Length of stay - ICU | From day of surgery until day of ICU stay.
  All patients will spend at least 1 day in the ICU for postoperative monitoring. ICU length of stay will be reported in days.
Length of stay - Hospital Discharge | From day of surgery until hospital discharge
  Hospital length of stay will be reported in days.

CONTACTS AND LOCATIONS:
Overall Officials: Vasileia Nyktari, MD,PhD, Study Chair — University of Crete, Medical School
Locations (1):
- University of Crete, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norman PE, Semmens JB, Lawrence-Brown MM. Long-term relative survival following surgery for abdominal aortic aneurysm: a review. Cardiovasc Surg. 2001 Jun;9(3):219-24. doi: 10.1016/s0967-2109(00)00126-5. PMID 11336844
- [Background] Johal AS, Loftus IM, Boyle JR, Heikkila K, Waton S, Cromwell DA. Long-term survival after endovascular and open repair of unruptured abdominal aortic aneurysm. Br J Surg. 2019 Dec;106(13):1784-1793. doi: 10.1002/bjs.11215. PMID 31747067
- [Background] Moris DN, Kontos MI, Mantonakis EI, Athanasiou AK, Spartalis ED, Bakoyiannis CN, Chrousos GP, Georgopoulos SE. Concept of the aortic aneurysm repair-related surgical stress: a review of the literature. Int J Clin Exp Med. 2014 Sep 15;7(9):2402-12. eCollection 2014. PMID 25356092
- [Background] Tsilimigras DI, Sigala F, Karaolanis G, Ntanasis-Stathopoulos I, Spartalis E, Spartalis M, Patelis N, Papalampros A, Long C, Moris D. Cytokines as biomarkers of inflammatory response after open versus endovascular repair of abdominal aortic aneurysms: a systematic review. Acta Pharmacol Sin. 2018 Jul;39(7):1164-1175. doi: 10.1038/aps.2017.212. Epub 2018 May 17. PMID 29770795
- [Background] Pearson S, Hassen T, Spark JI, Cabot J, Cowled P, Fitridge R. Endovascular repair of abdominal aortic aneurysm reduces intraoperative cortisol and perioperative morbidity. J Vasc Surg. 2005 Jun;41(6):919-25. doi: 10.1016/j.jvs.2005.02.040. PMID 15944585
- [Background] Wilt TJ, Lederle FA, Macdonald R, Jonk YC, Rector TS, Kane RL. Comparison of endovascular and open surgical repairs for abdominal aortic aneurysm. Evid Rep Technol Assess (Full Rep). 2006 Aug;(144):1-113. PMID 17764213
- [Background] Moore WS, Kashyap VS, Vescera CL, Quinones-Baldrich WJ. Abdominal aortic aneurysm: a 6-year comparison of endovascular versus transabdominal repair. Ann Surg. 1999 Sep;230(3):298-306; discussion 306-8. doi: 10.1097/00000658-199909000-00003. PMID 10493477
- [Background] Salartash K, Sternbergh WC 3rd, York JW, Money SR. Comparison of open transabdominal AAA repair with endovascular AAA repair in reduction of postoperative stress response. Ann Vasc Surg. 2001 Jan;15(1):53-9. doi: 10.1007/s100160010014. PMID 11221945
- [Background] Panaretou V, Siafaka I, Theodorou D, Manouras A, Seretis C, Gourgiotis S, Katsaragakis S, Sigala F, Zografos G, Filis K. Combined general-epidural anesthesia with continuous postoperative epidural analgesia preserves sigmoid colon perfusion in elective infrarenal aortic aneurysm repair. Saudi J Anaesth. 2012 Oct-Dec;6(4):373-9. doi: 10.4103/1658-354X.105870. PMID 23493852
- [Background] Jessula S, Atkinson L, Casey P, Kwofie K, Stewart S, Lee MS, Smith M, Herman CR. Surgically positioned paravertebral catheters and postoperative analgesia after open abdominal aortic aneurysm repair. J Vasc Surg. 2019 Nov;70(5):1479-1487. doi: 10.1016/j.jvs.2019.02.037. Epub 2019 May 29. PMID 31153699
- [Background] Panaretou V, Toufektzian L, Siafaka I, Kouroukli I, Sigala F, Vlachopoulos C, Katsaragakis S, Zografos G, Filis K. Postoperative pulmonary function after open abdominal aortic aneurysm repair in patients with chronic obstructive pulmonary disease: epidural versus intravenous analgesia. Ann Vasc Surg. 2012 Feb;26(2):149-55. doi: 10.1016/j.avsg.2011.04.009. Epub 2011 Oct 22. PMID 22018500
- [Background] Greco KJ, Brovman EY, Nguyen LL, Urman RD. The Impact of Epidural Analgesia on Perioperative Morbidity or Mortality after Open Abdominal Aortic Aneurysm Repair. Ann Vasc Surg. 2020 Jul;66:44-53. doi: 10.1016/j.avsg.2019.10.054. Epub 2019 Oct 28. PMID 31672606
- [Background] Ammar AS, Mahmoud KM. Comparative effect of propofol versus sevoflurane on renal ischemia/reperfusion injury after elective open abdominal aortic aneurysm repair. Saudi J Anaesth. 2016 Jul-Sep;10(3):301-7. doi: 10.4103/1658-354X.174907. PMID 27375385
- [Background] Loggi S, Mininno N, Damiani E, Marini B, Adrario E, Scorcella C, Domizi R, Carsetti A, Pantanetti S, Pagliariccio G, Carbonari L, Donati A. Changes in the sublingual microcirculation following aortic surgery under balanced or total intravenous anaesthesia: a prospective observational study. BMC Anesthesiol. 2019 Jan 5;19(1):1. doi: 10.1186/s12871-018-0673-7. PMID 30611197
- [Background] Giudice V, Lauwick S, Kaba A, Joris J. [Proven and expected benefits of intravenous lidocaine administered during the perioperative period]. Rev Med Liege. 2012 Feb;67(2):81-4. French. PMID 22482237
- [Background] Liu FL, Chen TL, Chen RM. Mechanisms of ketamine-induced immunosuppression. Acta Anaesthesiol Taiwan. 2012 Dec;50(4):172-7. doi: 10.1016/j.aat.2012.12.001. Epub 2013 Jan 11. PMID 23385040
- [Background] Mojtahedzadeh M, Chelkeba L, Ranjvar-Shahrivar M, Najafi A, Moini M, Najmeddin F, Sadeghi K, Barkhordari K, Gheymati A, Ahmadi A. Randomized Trial of the Effect of Magnesium Sulfate Continuous Infusion on IL-6 and CRP Serum Levels Following Abdominal Aortic Aneurysm Surgery. Iran J Pharm Res. 2016 Fall;15(4):951-956. PMID 28243294
- [Background] Marik PE. Propofol: an immunomodulating agent. Pharmacotherapy. 2005 May;25(5 Pt 2):28S-33S. doi: 10.1592/phco.2005.25.5_part_2.28s. PMID 15899746
- [Background] Roeckel LA, Utard V, Reiss D, Mouheiche J, Maurin H, Robe A, Audouard E, Wood JN, Goumon Y, Simonin F, Gaveriaux-Ruff C. Morphine-induced hyperalgesia involves mu opioid receptors and the metabolite morphine-3-glucuronide. Sci Rep. 2017 Sep 4;7(1):10406. doi: 10.1038/s41598-017-11120-4. PMID 28871199
- [Background] Yi P, Pryzbylkowski P. Opioid Induced Hyperalgesia. Pain Med. 2015 Oct;16 Suppl 1:S32-6. doi: 10.1111/pme.12914. PMID 26461074
- [Background] Mauermann E, Filitz J, Dolder P, Rentsch KM, Bandschapp O, Ruppen W. Does Fentanyl Lead to Opioid-induced Hyperalgesia in Healthy Volunteers?: A Double-blind, Randomized, Crossover Trial. Anesthesiology. 2016 Feb;124(2):453-63. doi: 10.1097/ALN.0000000000000976. PMID 26655493